CLINICAL TRIAL: NCT02415894
Title: Mifepristone and Misoprostol for Mid-trimester Termination of Pregnancy (13-22 Weeks LMP) in Ukraine
Brief Title: Mifepristone and Misoprostol for Mid-trimester Termination of Pregnancy in Ukraine
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Other Study IDs: 1025
Record Dates: First submitted 2015-04-02; First posted 2015-04-14 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Other Abortion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to examine the effectiveness and feasibility of a mifepristone-misoprostol medical abortion regimen in terminating pregnancies 13-22 weeks in Ukraine.

ELIGIBILITY:
Inclusion Criteria:

* Having an ongoing pregnancy of 13-22 weeks gestation
* Be willing to undergo surgical completion if necessary
* Have no contraindications to study procedures, according to provider
* Be willing and able to consent to participate in the study
* Be willing to follow study procedures

Exclusion Criteria:

* Known allergy to mifepristone or misoprostol/prostaglandin
* Any contraindications to vaginal delivery, including placenta previa
* Unable to provide consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women with mid-trimester pregnancy seeking abortion
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Rate of successful abortion | 15 hours after start of misoprostol induction

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Tsereteli, MD, PhD, Study Director — Gynuity Health Projects; Galina Maistruk, MD, Study Director — Woman Health and Family Planning Charitable Foundation
Locations (3):
- Ukraine (3):
  - Odessa Regional Hospital, Odesa
  - Poltava City Maternity Hospital, Poltava
  - Vinnitsa Regional Hospital, Vinnitsa

REFERENCES:
- [Derived] Platais I, Tsereteli T, Maystruk G, Kurbanbekova D, Winikoff B. A prospective study of mifepristone and unlimited dosing of sublingual misoprostol for termination of second-trimester pregnancy in Uzbekistan and Ukraine. BMJ Sex Reprod Health. 2019 Jun 4:bmjsrh-2018-200167. doi: 10.1136/bmjsrh-2018-200167. Online ahead of print. PMID 31164394